CLINICAL TRIAL: NCT06125717
Title: A Phase 1, Randomized, Rater and Subject Blinded Placebo Controlled Study to Evaluate the Safety, Reactogenicity, Tolerability and Immunogenicity of a Standard and a Fractional Dose of H1 Influenza Vaccine Delivered by VX-103 (a MIMIX Microneedle Patch (MAP) System) in Healthy Adults ≥18-39 Years of Age
Brief Title: Phase 1 Evaluation of H1 Influenza Vaccine Delivered by MIMIX MAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxess Technologies (Industry)
Collaborators: ICON plc (Industry); Q2 Solutions (Industry); Centricity Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: VX-103-01
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15 μg of the H1 influenza antigen (Active Comparator)
  Interventions: Biological: H1 influenza antigen
- 7.5 μg of the H1 influenza antigen (Active Comparator)
  Interventions: Biological: H1 influenza antigen
- Placebo (no antigen) (Placebo Comparator)
  Interventions: Biological: H1 influenza antigen

INTERVENTIONS:
Biological: H1 influenza antigen — Either 7.5 μg or 15 μg of the H1 influenza antigen

SUMMARY:
A Phase 1, Randomized, Rater and Participant Blinded Placebo Controlled Study to Evaluate the Safety, Reactogenicity, Tolerability and Immunogenicity of a Standard and a Fractional Dose of H1 Influenza Vaccine Delivered by VX-103 (a MIMIX Microneedle Array Patch (MAP) System) in Healthy Adults ≥18-39 Years of Age

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 39 years inclusive
* Provide written informed consent to participate
* Healthy participants without acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality

  o As determined by medical history, physical exam, laboratory screening
* Body Mass Index 18-35 kg/m2, inclusive, at screening

Exclusion Criteria:

* Any medical condition that in the judgement of the investigator would make subject participation in the study unsafe.
* Having cancer or received treatment for cancer within three years (persons with a history of cancer who are disease-free without treatment for three years or more are eligible), excluding basal cell carcinoma (BCC) or squamous cell carcinoma (SCC), which are allowed unless located at the vaccination site.
* Impaired immune responsiveness (of any cause), including diabetes mellitus.
* Receipt or plan to receive a non-study vaccine within 30 days prior to vaccination or 60 days after vaccination.
* Receipt of any influenza vaccine in previous 24 months and/or planned receipt of influenza vaccine for the duration of the study.
* Diagnosed influenza infection in the previous 24 months prior to screening.
* Diagnosed COVID infection via medical personnel or at home test within the past 60 days prior to screening
* Allergy to influenza vaccine or components, or history of severe local or systemic reaction to any vaccination.
* History of anaphylactic type reaction to injected vaccines
* History of or current allergy to latex
* History of Guillain-Barré Syndrome.
* Positive test result for hepatitis B surface antigen (HBsAg,), hepatitis C virus antibody (HBcAb), or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening.
* History of chronic obstructive pulmonary disease or history of other lung disease.
* History of severe allergic reactions to eggs.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
To determine the safety of VX-103 delivered as a single MIMIX MAP immunization | 180 Days

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Centricity Research Toronto, Toronto, Ontario
  - Centricity Research Mirabel, Mirabel, Quebec
  - Centricity Research Pointe-Claire, Pointe-Claire, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garg N, Tellier G, Vale N, Kluge J, Portman JL, Markowska A, Tussey L. Phase 1, randomized, rater and participant blinded placebo-controlled study of the safety, reactogenicity, tolerability and immunogenicity of H1N1 influenza vaccine delivered by VX-103 (a MIMIX microneedle patch [MAP] system) in healthy adults. PLoS One. 2024 Jun 6;19(6):e0303450. doi: 10.1371/journal.pone.0303450. eCollection 2024. PMID 38843267